CLINICAL TRIAL: NCT00296725
Title: Dichotic Listening as a Predictor of Placebo and Medication Response in Depression
Brief Title: Dichotic Listening as a Predictor of Medication Response in Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jonathan W Stewart, M.D, Clinical Psychiatrist, New York State Psychiatric Institute
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: #4217R/#5294R; continuation of IRB3112; (Other Grant/Funding Number: There is no grantor or funder); became IRB5294R. (Other Grant/Funding Number: there is no grantor or funder)
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Major Depression; Dysthymia; Depressive Disorder Not Otherwise Specified
Keywords: Major Depression; Dysthymia; Depression Not Otherwise Specified; Dichotic Listening; Fluoxetine; Imipramine; Predictors
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Fluoxetine; Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluoxetine / Imipramine (Experimental): fluoxetine or Imipramine
  Interventions: Drug: Fluoxetine; Drug: Imipramine

INTERVENTIONS:
Drug: Fluoxetine — Phase 1: Fluoxetine: wk 1: 10 mg/day; wks 2-3: 20 mg/day; wks 4-5: 40 mg/day; wk 6: 60 mg/day; wks 7-12: 80 mg/day *All increases only if tolerated.
  Other Names: Prozac
Drug: Imipramine — Phase 2: Imipramine wk 1: 25 mg/day; wk 2: 50 mg/day; wk 3: 100 mg/day, 150 mg/day after 3 days; wk 4: 200 mg/day, 250 mg/day after 3 days; wks 5-6: 300 mg/day. *All increases only if tolerated.
  Other Names: Tofranil

SUMMARY:
Depressed patients will have hearing tests and then be treated with up to three treatments (i.e., Fluoxetine, Imipramine) until remitted, to see whether test results predict specific outcomes.

DETAILED DESCRIPTION:
100 depressed patients will be tested with verbal and nonverbal dichotic tests, and then treated sequentially with Fluoxetine and Imipramine until remitted. Preferential hemisphere for auditory processing will be correlated with treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-65
* Meets Diagnostic and Statistical Manual, 4th Edition criteria for current Major Depression, Dysthymia or Depression Not Otherwise Specified

Exclusion Criteria:

* Known hearing impairment
* Active suicidal ideation (history of suicide attempts will be evaluated on a case by case basis)
* Hamilton Rating Scale for Depression, 17-item version > 20
* Current (past six months) alcohol and/or drug abuse or dependence
* Medical condition likely to require intervention contraindicated with study medication (e.g., known arrhythmia likely to be exacerbated by Imipramine)
* Bipolar I
* Psychosis
* If currently taking antidepressants or mood stabilizers, cannot be off psychotropic medication for 7 weeks (10 weeks for Prozac) or felt to require other psychiatric medication (other than occasional sleep or Anxiety medication)
* Premenopausal women not using known effective birth control
* Not currently depressed (whether considered due to current treatment or not)
* Nonresponse to adequate trial of both study medications (i.e., > 4weeks on > escitalopram 30 mg/d, and imipramine 200 mg/d); patients having an inadequate response to one study medication could be enrolled and receive the other; patients having responded to an adequate trial of either study medication would be offered a retrial; also excluded will be subjects having non responded to an adequate trial with citalopram (i.e., > 4 weeks on > citalopram 60 mg/d)
* Left-handed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1994-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, MD., Principal Investigator — New York State Psychiatric Institute - Columbia University Department of Psychiatry
Locations (1):
- Depression Evaluation Service, New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Bruder GE, Otto MW, McGrath PJ, Stewart JW, Fava M, Rosenbaum JF, Quitkin FM. Dichotic listening before and after fluoxetine treatment for major depression: relations of laterality to therapeutic response. Neuropsychopharmacology. 1996 Aug;15(2):171-9. doi: 10.1016/0893-133X(95)00180-L. PMID 8840353
- [Background] Bruder GE, Stewart JW, Tenke CE, McGrath PJ, Leite P, Bhattacharya N, Quitkin FM. Electroencephalographic and perceptual asymmetry differences between responders and nonresponders to an SSRI antidepressant. Biol Psychiatry. 2001 Mar 1;49(5):416-25. doi: 10.1016/s0006-3223(00)01016-7. PMID 11274653
- [Background] Bruder GE, Stewart JW, McGrath PJ, Deliyannides D, Quitkin FM. Dichotic listening tests of functional brain asymmetry predict response to fluoxetine in depressed women and men. Neuropsychopharmacology. 2004 Sep;29(9):1752-61. doi: 10.1038/sj.npp.1300519. PMID 15238992
- [Background] Stewart JW, Quitkin FM, McGrath PJ, Bruder GE. Do tricyclic responders have different brain laterality? J Abnorm Psychol. 1999 Nov;108(4):707-10. doi: 10.1037//0021-843x.108.4.707. PMID 10609436
- [Background] Bruder GE, Stewart JW, Voglmaier MM, Harrison WM, McGrath P, Tricamo E, Quitkin FM. Cerebral laterality and depression: relations of perceptual asymmetry to outcome of treatment with tricyclic antidepressants. Neuropsychopharmacology. 1990 Feb;3(1):1-10. PMID 2306330
- [Derived] Bruder GE, Sedoruk JP, Stewart JW, McGrath PJ, Quitkin FM, Tenke CE. Electroencephalographic alpha measures predict therapeutic response to a selective serotonin reuptake inhibitor antidepressant: pre- and post-treatment findings. Biol Psychiatry. 2008 Jun 15;63(12):1171-7. doi: 10.1016/j.biopsych.2007.10.009. Epub 2007 Dec 3. PMID 18061147
- See also: Depression Evaluation Service - official website — http://www.depression-nyc.org
- See also: New York State Psychiatric Institute - official website — http://www.nyspi.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 Screened. 4 did not return, 2 withdrew consent. Period 1 started with 17 participants available and eligible to participate in period I were treated with fluoxetine; 2 fluoxetine non-responders, 3 non-remiiters and 3/5 dropouts (n=8) continued to Period 2.
Pre-assignment Details: 17 participants available and eligible to participate in period I
Groups:
- Fluoxetine / Imipramine: Fluoxetine: wk 1: 10 mg/day; wks 2-3: 20 mg/day; wks 4-5: 40 mg/day; wk 6: 60 mg/day; wks 7-12: 80 mg/day *All increases only if tolerated.
  Imipramine: wk 1: 25 mg/day; wk 2: 50 mg/day; wk 3: 100 mg/day, 150 mg/day after 3 days; wk 4: 200 mg/day, 250 mg/day after 3 days; wks 5-6: 300 mg/day. *All increases only if tolerated.
Period: Phase 1: Fluoxetine (1-12 Weeks)
Arm/Group | Fluoxetine / Imipramine
Started (Follow reviewers suggestion, added 2 periods to avoid double counting. Period 1 started with 17) | 17
Completed | 12
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 4
Period: Phase 2: Imipramine (1-6 Weeks)
Arm/Group | Fluoxetine / Imipramine
Started (8 participants available and eligible to participate in period 2) | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline data collected for all 25 enrolled participants
Arm/Group | Fluoxetine / Imipramine
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years as reported by subject
  years | 37 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Scale (HAM-D)
Description: The HAM-D is a commonly used measure of the severity of depression. While several versions exist consisting of different numbers of items, virtually all include the original 17. Each item is scored from on a 3 or 5 point scale (so, from 0-2 or 0-4), with 0 indicating the item is not present and the highest item score indicating it is present nearly all the time to the severest extent. Item scores are added to obtain a total HAM-D score. Minimum possible score is 0 (indicating none of the 17 items is present), maximal possible score is 52. By convention, scores of <=7 are accepted as indicating "remission" and scores that have decreased >= 50% from pre-treatment indicate positive "response". Higher scores indicate worse depression, while lower scores indicate milder depression or lack of depressive symptoms.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fluoxetine: fluoxetine
  Fluoxetine: wk 1: 10 mg/day; wks 2-3: 20 mg/day; wks 4-5: 40 mg/day; wk 6: 60 mg/day; wks 7-12: 80 mg/day *All increases only if tolerated.
- Imipramine: imipramine
  Imipramine: wk 1: 25 mg/day; wk 2: 50 mg/day; wk 3: 100 mg/day, 150 mg/day after 3 days; wk 4: 200 mg/day, 250 mg/day after 3 days; wks 5-6: 300 mg/day. *All increases only if tolerated.
Arm/Group | Fluoxetine | Imipramine
Number analyzed (Participants) | 17 | 8
score on a scale | 10 (7) | 9 (7)

2. Secondary Outcome: Number of Participants With Positive Response as Assessed by the Clinical Global Impression -Global Improvement Scale (CGI-I)
Description: The CGI consists of two ratings: 1) Global Severity (CGI-S) and 2) Global Improvement (CGI-I), both having seven possible ratings, each from 1-7. Ratings on the CGI-S are: 1="No psychopathology" 2="Minimal psychopathology" 3="Mild psychopathology 4="Moderate psychopathology" 5="Moderately severe psychopathology" 6="Severe psychopathology" 7 "Extreme psychopathology". CGI-I ratings are rated for how the past week's psychopathology compares to the week immediately prior to start of treatment and includes: 1="Very much improved" 2="much improved" 3="minimally improved" 4="Unchanged" 5="minimally worse" 6="much worse" 7="very much worse". Scores on both thus range from 1-7 with lower scores indicating less psychopathology/greater improvement, respectively, and higher scores indicating more psychopathology/less improvement, respectively. We define "response" as a CGI-I of 1 or 2; "nonresponse" is all other ratings (i.e., CGI-I = 3 or higher.
Time Frame: 6 weeks.
Population: Response Rate
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoxetine | Imipramine
Number analyzed (Participants) | 17 | 8
Participants | 7 | 4

ADVERSE EVENTS:
Arm/Group | Fluoxetine | Imipramine
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/8
Other Adverse Events (participants affected / at risk) | 7/17 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=17) | Imipramine (N=8)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — feeling short of breath
irritability (Psychiatric disorders) | 1 (1) | 0 (0) — patient reports feeling irritable
rash (Immune system disorders) | 2 (2) | 0 (0) — urticaria
lost to follow-up (General disorders) | 3 (3) | 1 (1) — Patient did not return for regular visits and did not respond to telephone messages or letters

LIMITATIONS AND CAVEATS:
Open, non-randomized treatment and ratings; small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No